CLINICAL TRIAL: NCT07365150
Title: PRECISion usE of TRANexamic Acid for Supratentorial Acute Cerebral Hemorrhage Trial: a Pilot Randomized Controlled Trial
Brief Title: Precision Use of TXA in Intracerebral Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Kong Kong (Unknown); Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Teo Kay-Cheong, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TKC202403
Record Dates: First submitted 2026-01-02; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Intracerebral Hemorrhage
Keywords: Tranexamic acid; Intracerebral hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial with PROBE design
Who Masked: Outcomes Assessor
Masking Description: Assessor of clinical outcomes (GCS, NIHSS and mRS) and hematoma volume will be blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXA arm (Active Comparator): TXA 1000mg stat over 10 minutes and 1000 mg over 8 hours
  Interventions: Drug: Tranexamic Acid (IV)
- Control arm (No Intervention): No TXA

INTERVENTIONS:
Drug: Tranexamic Acid (IV) — TXA 1000mg stat over 10 minutes and 1000 mg over 8 hours
  Arms: TXA arm

SUMMARY:
Primary Intracerebral hemorrhage (ICH) is a severe and disabling disease. The hematoma will expand within the first few hours, which contributes to increasing brain injury and worsening neurological prognosis. Hence, one of ICH's main acute therapeutic strategies is to reduce hematoma expansion (HE) with hemostatic agents like tranexamic acid (TXA) or recombinant factor VIIa. However, although most HE trials have demonstrated that treatment attenuated HE, they have largely been unable to demonstrate therapeutic benefit in improving functional outcomes. The lack of outcome benefits for ICH treatment is because therapeutic benefits are significantly confounded by the outcome heterogeneity based on ICH location and the variation in the degree of HE between patients, which is not accounted for in all ICH trials.

The investigators' recent work has examined the interplay between ICH location and volume in determining ICH pathophysiology and outcomes, highlighting a critical interaction between these factors and neurological prognosis. Also, as HE only occurs in 15-40% of patients, the therapeutic benefits of treatment targeting HE are not modifiable in most patients. Furthermore, only a minority of patients with HE experienced neurological deterioration (HE-related neurological deterioration) that could impact their neurological outcomes. There is also a location-specific variation in the risk of HE-related neurological deterioration, occurring at a larger baseline volume for ICH at putamen/ lobar compared to thalamus/ internal capsule. Hence, as outcome heterogeneity based on ICH location and the variation in the degree of HE significantly confounds therapeutic effect, better patient selection for hemostatic agents in ICH treatment is essential to yield functional benefit.

To address this, a novel selection criteria (>7ml for thalamus/ internal capsule, >30ml for putamen/ lobar) is proposed, which, in theory, would account for the confounding effect of location-specific outcome heterogeneity and the location-based variation in HE-related neurological deterioration. Therefore, the PRECISE-TRANSACT trial aims to investigate whether TXA administration based on this selection criteria significantly reduces the risk of neurological deterioration and consequent therapeutic benefit.

ELIGIBILITY:
Inclusion Criteria:

* Primary ICH Diagnosis
* Age ≥ 18 years
* Within 6 hours of ICH
* Supratentorial ICH
* GCS ≥8
* Location-specific volume criteria (>7ml for thalamus or internal capsule; >30ml for putamen or lobar)

Exclusion Criteria:

* Severe pre-morbid disability (Pre-morbid modified Rankin scale 5)
* Anticipated surgical treatment
* Recent acute atherosclerotic cardiovascular diseases (e.g. acute coronary syndrome, ischemic stroke)
* Receiving anticoagulation
* Recent intravascular stent placement and on dual antiplatelet treatment
* Expected life expectancy of <1 year
* Inability to participate in follow-up activity
* Bleeding tendency
* Severe renal impairment
* Severe liver impairment
* Known contraindication or allergy to tranexamic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Trial recruitment rate | At recruitment
  Number of patients recruited per month
Trial retention rate | Six months
  Number of patients who completed follow-up

SECONDARY OUTCOMES:
The number of patients with early neurological deterioration | 24 hours of admission
  Early neurological deterioration is defined as ≥4-point increase in the National Institute of Health Stroke Scale (NIHSS) or ≥2-point decrease in the Glasgow Coma Scale (GCS) within 24 hours
The number of patients with delayed neurological deterioration or any deterioration | Day 2-7
  1. Delayed neurological deterioration is defined as ≥4-point increase in the NIHSS or ≥2-point decrease in the GCS within day 2-7.
  2. Any deterioration is defined as any deterioration in NIHSS, GCS, or limb power grade within 7 days.
Modified Rankin Scale | Six months
  Neurological recovery will be assessed using the Modified Rankin Scale (mRS), which ranges from 0 to 6, where 0 indicates no symptoms, 1-5 indicate increasing levels of neurological disability, and 6 indicates death.
Hematoma expansion | 24 hours
  Increase in hematoma volume from baseline to reassessment imaging

OTHER OUTCOMES:
Thrombotic event | 30 days
  Any arterial or venous thrombotic events.
Mortality | 30 days
  All caused death

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong